CLINICAL TRIAL: NCT03189836
Title: Phase 1 Study of ACTR707, an Autologous T Cell Product, in Combination With Rituximab, in Subjects With Relapsed or Refractory CD20+ B Cell Lymphoma
Brief Title: Study of ACTR707 in Combination With Rituximab in Subjects With Relapsed or Refractory B Cell Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision
Sponsor: Cogent Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATTCK-20-03
Record Dates: First submitted 2017-06-12; First posted 2017-06-16 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Lymphoma
Keywords: CD20+; B cell; ACTR; ACTR707; relapsed; refractory; T cell; T cell product; adoptive T cells; gene therapy
MeSH Terms: conditions — Lymphoma; Recurrence | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ACTR707 in combination with rituximab (Experimental)
  Interventions: Biological: ACTR707; Biological: rituximab

INTERVENTIONS:
Biological: ACTR707 — autologous T cell product
Biological: rituximab — CD20-directed cytolytic antibody

SUMMARY:
This is a phase 1, multi-center, single-arm, open-label study evaluating the safety and anti-lymphoma activity of an autologous T cell product (ACTR707) in combination with rituximab in subjects with refractory or relapsed CD20+ B cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* signed written informed consent obtained prior to study procedures
* histologically-confirmed relapsed or refractory CD20+ B-cell lymphoma of one of the following types, with documented disease progression or recurrence following the immediate prior therapy: DLBCL (regardless of cell of origin or underlying molecular genetics), MCL, PMBCL, Gr3b-FL, TH-FL (prior dx of FL before transforming to DLBCL).
* biopsy-confirmed CD20+ expression of the underlying malignancy with disease progression following immediate prior therapy
* at least 1 measurable lesion on imaging.
* must have received adequate prior therapy for the underlying CD20+ B-cell lymphoma, defined as an anti-CD20 mAb in combination with an anthracycline-containing chemotherapy regimen (i.e. chemo-immunotherapy) and at least one of the following:

  * biopsy-proven refractory disease after frontline chemo-immunotherapy
  * relapse within 1 year from frontline chemo-immunotherapy and ineligible for autologous hematopoietic stem cell transplant (auto-HSCT)
  * for subjects with DLBCL, PMBCL, and Gr3b-FL: relapsed or refractory disease following at least 2 prior regimens or following an auto-HSCT
  * for subjects with TH-FL: relapsed or refractory disease following at least 2 prior regimens or following an auto-HSCT. At least 1 prior regimen with an anti-CD20 mAb in combination with chemotherapy is required following documented transformation
  * for subjects with MCL (confirmed with cyclin D1 expression or evidence of t(11;14) by cytogenetics, fluorescent in situ hybridization (FISH) or polymerase chain reaction (PCR): relapsed or refractory disease after at least 1 prior regimen with chemo-immunotherapy (prior auto-HSCT is allowable)
* ECOG 0 or 1
* life expectancy of at least 6 months
* platelet count greater than 50,000/µL

Exclusion Criteria:

* known active central nervous system (CNS) involvement by malignancy.
* prior treatment as follows:

  * alemtuzumab within 6 months of enrollment
  * fludarabine, cladribine, or clofarabine within 3 months of enrollment
  * external beam radiation within 2 weeks of enrollment
  * mAb (including rituximab) within 2 weeks of enrollment
  * other lymphotoxic chemotherapy (including steroids except as below) within 2 weeks of enrollment
  * experimental agents within 3 half-lives prior to enrollment, unless progression is documented on therapy
* clinically significant cardiac disease
* clinically significant active infection
* clinically significant CNS disorder
* clinical history, prior diagnosis, or overt evidence of autoimmune disease
* known bone marrow involvement due to underlying malignant disease, in dose-escalation phase only

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-10-04 (Actual); Primary Completion 2020-09-21 (Actual); Study Completion 2020-09-21 (Actual)

PRIMARY OUTCOMES:
Safety as assessed by dose limiting toxicities (DLTs) | 28 days
  Dose-limiting toxicities, MTD, incidence and severity of AEs and clinically significant abnormalities of laboratory values
Determination of maximum tolerated dose and proposed recommended Phase 2 dose | 24 weeks

SECONDARY OUTCOMES:
Anti-lymphoma activity as measured by overall response rate | 24 weeks
Anti-lymphoma activity as measured by duration of response | 24 weeks
Anti-lymphoma activity as measured by progression-free survival | 24 weeks
Anti-lymphoma activity as measure by overall survival | 24 weeks
Assessment of persistence of ACTR707 as measured by flow cytometry and qPCR | 24 weeks
Assessment of ACTR707 phenotype and function as measured by flow cytometry | 24 weeks
Assessment of inflammatory markers and cytokines/chemokines | 24 weeks
  Cytokines and Inflammatory markers
Rituximab PK | 24 weeks
  Rituximab plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Sachs, MD, Study Director — Cogent Biosciences, Inc.
Locations (11):
- United States (11):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Yale University, New Haven, Connecticut
  - Emory University, Winship Cancer Institute, Atlanta, Georgia
  - Loyola University, Maywood, Illinois
  - Indiana Bone and Marrow Transplantation, Indianapolis, Indiana
  - University of Maryland, Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - Ohio State University, Columbus, Ohio
  - Tennessee Oncology - Nashville, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338